CLINICAL TRIAL: NCT05736237
Title: Identification and Verification of Candidate Genes Responsible for Optic Disc Drusen
Brief Title: Identification and Verification of Candidate Genes Responsible for Optic Disc Drusen Development
Acronym: GENODD
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Alvilda Steensberg, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-20027930
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Optic Disk Drusen
Keywords: Optic disc drusen; Genetics
MeSH Terms: conditions — Optic Disk Drusen | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Families with optic disc drusen
  Interventions: Genetic: Whole exome sequencing

INTERVENTIONS:
Genetic: Whole exome sequencing — With Next Generation Sequenzing

SUMMARY:
The goal of this observational study is to learn about the genetic background for the development of optic disc drusen. The main question is:

• Can one or more candidate genes be found?

Participants will have a blood sample taken and answer a questionnaire.

DETAILED DESCRIPTION:
The study is an international collaboration between University of Utah, University of Sydney, University of Valladolid, and University of Copenhagen. Patients with Optic disc drusen from 15 known optic disc drusen-families from different countries (USA, Australia, Spain and Denmark) are participating in this study.

Blood samples are drawn from each patient and their affected and unaffected family members, and DNA will be extracted. The investigators will do an Optical coherence tomography-scan (according to ODDS Consortium guidelines), and the participant will be asked to fill out the Visual Function Questionnaire (VFQ-25) including four additional questions about optic disc drusen.

The etiology of optic disc drusen will be analyzed with a Whole Exome Sequencing (WES), with the use of Next Generation Sequencing (NGS). Prior to WES, all participants will receive genetic counseling by a consultant to ensure awareness of possible secondary genetic findings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18, who are capable of giving consent
* Diagnosis of optic disc drusen and a minimum of 3 optic disc drusen-affected family members

Exclusion Criteria:

* Less than 3 affected family members
* Under the age of 18 or mentally disabled

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Families with ODD
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Candidate gene | 2023-2024
  Genetics variants shared by the families will be compared with findings in the remaining families and identical genes will undergo further analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with the project responsible unit